CLINICAL TRIAL: NCT02614924
Title: Comparison of Flexible Fibreoptic Scope With Pentax AWS Videolaryngoscope for Ease of Intubation During Awake Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RD098211
Record Dates: First submitted 2015-11-24; First posted 2015-11-25 (Estimated); Results first posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Anesthesia Intubation Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flexible fibre-optic scope (Other): Randomly allocated to fibreoptic group
  Interventions: Device: Flexible fibreoptic scope; Device: Pentax AWS videolaryngoscope
- Pentax AWS videolaryngoscope (Other): Randomly allocated Pentax AWS videolaryngoscope
  Interventions: Device: Flexible fibreoptic scope; Device: Pentax AWS videolaryngoscope

INTERVENTIONS:
Device: Flexible fibreoptic scope — Patient intubated using fibreoptic scope
Device: Pentax AWS videolaryngoscope — Patient intubated using Pentax AWS videolaryngoscope

SUMMARY:
The purpose of this study is to identify whether Pentax Airway Scope (AWS) videolaryngoscope would be a more effective device compared to flexible fibreoptic scope (FOS) for awake intubation in a difficult airway.

DETAILED DESCRIPTION:
Background:

The incidence of difficult tracheal intubation during routine anaesthesia in general population is around 3-18% although it varies [1]. Awake intubation is considered in situations such as in patients with a known or suspected difficult airway, upper airway obstruction. Awake intubation under local anaesthesia and sedation also indicated cervical spine disease in view of minimising movement of cervical spine [2]. Any technique tracheal intubation under general anaesthesia involves some degree of movement at cervical spine. Direct laryngoscopy and tracheal intubation in under general anaesthesia is usually achieved by flexion of lower cervical spine and extension at atlanto-occipital joint [3]. Difficulties or failure in airway management is still an important factor in morbidity and mortality related to anaesthesia.

In recent years videolaryngoscopes have been used as an alternative to traditional fibreoptic scope in the management of difficult airway [4,7,8]. Over last 2 years in our institution the investigators have used Pentax AWS videolaryngoscope for awake intubation in patients presenting for surgery with cervical spine disease [9, 10].

However there has not been any study comparing flexible fibreoptic scope with video laryngoscopes in the management of difficult airway in awake patients. The proposed benefits of Pentax AWS (Airway scope) over a flexible fibreoptic scope include ease of setting up the device, less complexity of the skill, therefore easy to learn the skill and availability of disposable devices minimising the need for cleaning and disinfecting the device.

Pentax AWS with PBlade videolaryngoscope has a unique target symbol displayed on the monitor, which highlights the intended path of the endotracheal tube. The Pentax PBlade is a single patient use device that minimizes the risk of infection.

Study Design and Methods: Randomised Controlled Trial

Patient Selection:

Forty patients presenting for cervical spine surgery under general anaesthesia and requiring oral endotracheal intubation will be invited to take part in the study. During preoperative visit, a patient information sheet will be given to the patients meeting the eligible criteria. The patient will be given adequate time to read the information sheet and any queries will be answered. Wherever possible, suitable patients will be identified in the preoperative assessment clinic. A detailed airway assessment will be performed by one of the investigator.

Whenever possible, when patients are admitted the night before their operation, they should be seen by an Anaesthetist and given the study information.

Techniques of Anaesthesia:

After securing intravenous cannulation and instituting standard anaesthetic monitoring with ECG, pulse oximetry and non-invasive blood pressure monitoring, conscious sedation will be started using target controlled infusion of remifentanil and 1 mg of midazolam. At this stage numbered opaque envelope will be opened to choose one of the two devices. The tongue, oropharynx and larynx will be anaesthetised using 4% lignocaine using Mckenzie technique (nebulisation of local anaesthetic through 20 G cannula).

Adequate anaesthesia of upper airway will be checked by inserting an appropriately sized oropharyngeal airway (if the patient can tolerate well, the airway is anesthetised adequately, if not further local anaesthetic is administered to the oropharynx). After confirming adequate anaesthesia of upper airway, the chosen device will be inserted into the oropharynx. Further local anaesthesia to the base of the tongue, larynx and trachea will be administered using spray as you go technique where the local anaesthetic administered through the device whilst gradually advancing the device towards larynx. After confirming the position of the tracheal tube and testing the gross neurological state of all 4 limbs, general anaesthesia will be induced.

Data Collection:

During the procedure of laryngoscopy and endotracheal intubation, a modified intubation difficulty score (IDS) would be developed based on the parameter recorded. Along with intubation difficulty score other parameters compared include: time taken to complete the process of intubation, anaesthetist rating of intubation and patient rating of procedure.

The following parameter would be recorded and scored:

1. Coughing episode: 0 no cough 1 if mild cough, 2 if moderate cough, 3 if severe cough.
2. Gagging episode: 0 no gagging, 1 if mild gag, 2 if moderate gag, 3 if severe gag.
3. Ease of insertion of device: 0 easy, 1 if mild difficulty 2 if moderately difficulty, 3 very difficult.
4. Laryngoscope view based on the percentage of the glottis visualised 0 if 75-100% view, 1 if 50-75% view, 2 if <50% view, 3 no VC visible.
5. Tube rotation or manipulation, 0 if no rotation required, 1 if rotation required
6. Airway trauma, 0 no trauma, 1 if minor injury (lip), 2 if oro-pharyngeal injury/ bleeding. 3, bleeding requiring use of suction
7. Stress response based on heart rate and blood pressure (0 if stable, 1 if increased more than 20%)
8. Overall patients' tolerance as judged by the Anaesthetists (visual analogue score of 0 to 100mm)
9. Overall impression from patient on a visual analogue scale (visual analogue score of 0 to 100mm)

ELIGIBILITY:
Inclusion Criteria:

* Patients with cervical spine disease presenting for cervical spinal surgery and requiring awake intubation under local anaesthesia and conscious sedation.
* Patients with anticipated difficult airway include those with Mallampati class 3 and above, other signs such as limited neck movement and limited jaw protrusion will be include in the study

Exclusion Criteria:

* Children below 18 years of age, pregnant mothers and patients presenting with airway pathology will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between 27.11.12 till 24.7.14. Recruitment was done during anaesthetic prep assessment.
Pre-assignment Details: No participants were excluded
Groups:
- Pentax AWS Videolaryngoscope: Randomly allocated to Pentax AWS
Period: Overall Study
Arm/Group | Flexible Fibre-optic Scope | Pentax AWS Videolaryngoscope
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pentax AWS Videolaryngoscope Group: Randomly allocated Pentax AWS videolaryngoscope and intubated using Pentax AWS videolaryngoscope
- Total: Total of all reporting groups
Arm/Group | Flexible Fibre-optic Scope | Pentax AWS Videolaryngoscope Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 9 | 25
  >=65 years | 4 | 11 | 15
Age, Continuous [Median (Full Range); unit: years] | 55.5 [23 to 77] | 66.5 [44 to 77] | 60.5 [23 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 11 | 8 | 19
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Total Time Taken to Complete the Procedure of Awake Intubation
Time Frame: up to 20 minutes
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Flexible Fibre-optic Scope | Pentax AWS Videolaryngoscope
Number analyzed (Participants) | 20 | 20
seconds | 900 [739 to 1059] | 651 [601 to 720]

2. Secondary Outcome: Intubation Time
Time Frame: up to 10 minutes
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Flexible Fibre-optic Scope | Pentax AWS Videolaryngoscope
Number analyzed (Participants) | 20 | 20
seconds | 420 [283 to 480] | 183 [144 to 220]

ADVERSE EVENTS:
Time Frame: 20 months
Groups:
- Pentax AWS Videolaryngoscope: Randomly allocated to Pentax AWS group Pentax AWS videolaryngoscope group: Patient intubated with Pentax AWS
Arm/Group | Flexible Fibre-optic Scope | Pentax AWS Videolaryngoscope
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes